CLINICAL TRIAL: NCT05155540
Title: A Comparative Study of The Efficacy and Safety of Direct Mechanical Thrombectomy Versus Bridging Therapy in Large Vessel Occlusion: An Egyptian Single-Center Experience
Brief Title: Direct Mechanical Thrombectomy Versus Bridging Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Anwar, Principal Investigator, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201218
Record Dates: First submitted 2021-12-03; First posted 2021-12-13 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Thrombectomy; Ischemic Stroke; Large-Artery Atherosclerosis (Embolus/Thrombosis)
Keywords: ischemic stroke; Direct mechanical thrombectomy; Bridging therapy
MeSH Terms: conditions — Ischemic Stroke; Embolism; Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, prospective, double-arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Direct mechanical thrombectomy (Active Comparator): Direct mechanical thrombectomy performed within 4.5 of stroke onset without giving intravenous recombinant tissue plasminogen activator.
  Interventions: Device: Trevo and or Merci devices for stent retreival; Device: Penumbra system for stent aspiration
- Bridging therapy (Active Comparator): Mechanical thrombectomy performed within 4.5 of stroke onset after giving intravenous recombinant tissue plasminogen activator at a dose of 0.9 mg/Kg
  Interventions: Device: Trevo and or Merci devices for stent retreival; Device: Penumbra system for stent aspiration; Drug: recombinant tissue plasminogen activator

INTERVENTIONS:
Device: Trevo and or Merci devices for stent retreival — FDA approved devices for stent retrieval during mechanical thrombectomy
  Other Names: No other names
Device: Penumbra system for stent aspiration — FDA approved devices for stent aspiration during mechanical thrombectomy
Drug: recombinant tissue plasminogen activator — FDA approved drug for treatment of acute ischemic stroke within 4.5 hours of strokeonset
  Arms: Bridging therapy

SUMMARY:
This study compares the efficacy and safety of direct mechanical thrombectomy versus bridging therapy in patients with anterior circulation large vessel occlusion in a cohort of patients treated at the stroke unit of a single centre at Alexandria University in Egypt.

DETAILED DESCRIPTION:
This study compares the efficacy and safety of direct mechanical thrombectomy versus bridging therapy in patients with anterior circulation large vessel occlusion in a cohort of patients treated at the stroke unit of a single centre at Alexandria University in Egypt. In the first arm, 17 patients were recruited and underwent direct mechanical thrombectomy without receiving recombinant tissue plasminogen activator. In the bridging therapy arm, 34 patients received first tissue plasminogen activator then underwent direct mechanical thrombectomy. The efficacy was evaluated by the NIHSS improvement 24 hours following stroke onset and the modified Rankin scale 3 months following stroke. Safety was assessed by the procedural complications rate especially the hemorhagic transformation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior ischemic stroke due to large vessel occlusion.
* A previous autonomous modified Rankin Scale (mRS) of less than 2.
* A National Institutes of Health Stroke Scale (NIHSS)≥4
* A groin puncture within 4.5 hours of the neurological deficit onset.

Exclusion Criteria:

* Imaging documentation of intracranial haemorrhage
* A premorbid mRS score of 2 or more
* Absence of diffusion perfusion mismatch in CT perfusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 3 months
  A measurement of functional independence following ischemic stroke
Complication rate | within one week postoperatively
  The rate and type of complications occuring postoperatively

SECONDARY OUTCOMES:
The National Institutes of Health Stroke Scale (NIHSS) score | at 24 hours postoperatively
  A validated scale for assessment of neurological dysfunction associated with stroke

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Abdel Ghani, Master's, Principal Investigator — Alexandria University Faculty of Medicine
Locations (1):
- Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon request
Supporting Information: Study Protocol, SAP
Time Frame: 30 days
Access Criteria: The data will be available upon request